CLINICAL TRIAL: NCT02706002
Title: Fluoroscopy Improves Femoral Stem Placement in Cementless Total Hip Arthroplasty
Brief Title: Fluoroscopy Improves Femoral Stem Placement
Acronym: Fluoroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Haluk Çabuk, MD, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OkmeydaniTRH
Record Dates: First submitted 2016-02-25; First posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Fluoroscopy; Hip Prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hip prosthesis under fluoroscopy (Active Comparator): implantation of femoral stem of hip prosthesis in this group of patients are under fluoroscopic guidance for stem size and stem alignment and last rap before original stem implantation will be checked for alignment , lateral and vertical offsets parameters.
  Interventions: Device: fluoroscopy; Procedure: hip prosthesis
- hip prosthesis without fluoroscopy (Sham Comparator): in this group of patients rasping of femoral canal during hip prosthesis is made via anatomic landmarks which confirmed by to senior surgeons and than original stem implanted.
  Interventions: Procedure: hip prosthesis

INTERVENTIONS:
Device: fluoroscopy — in active group femural stem of hip prosthesis will implanted under fluoroscopy guidance during operation till maximum rasp size reached that fills the medullary canal. ordinary 3-5 sequences per operation
  Arms: hip prosthesis under fluoroscopy
Procedure: hip prosthesis — all patients in the study will undergo hip prosthesis

SUMMARY:
Fluoroscopy is routinely used in trauma cases to evaluate alignment and reduction quality. Because conventional templating has a high mismatch rate, the investigators sought to explore whether the investigators could use intraoperative fluoroscopy while implanting the femoral stem.

DETAILED DESCRIPTION:
Prospectively two groups of patients with hip osteoarthritis were included in the study. Hip osteoarthritis was classified according to the Croft classification. The investigators primary goal is to evaluate T+ 2 ( 2 cm above trochanter minor) results between the two groups. Standard effect sizes (standard effect size) assumed to be at least 0.75. 30 cases for each group took power with 80% margin of 5% error. Patients with malignant tumors, previously known bone disease, drug consumption affecting bone mineralization or Crowe type III hip dislocations with greater than 4 cm of limb length discrepancy (LLD) were excluded. Prior to the operation, all patients underwent an X ray investigation to exclude any bone abnormalities. All patients were operated by the same team, which was composed of two senior surgeons and 2 fellows. Patients with odd-numbered were the first group and even numbers were the second group in order of receipt surgery. All patients were operated on the lateral decubitus position with a posterior approach and a metaphyseal locking femoral stem (Depuy Synthess SUMMIT Tapered Hip System, US). In the first group, no preoperative templating was performed, and the final conformation of the stem size and position was decided freehand intraoperatively based on anatomic landmarks. In the second group, there was also no preoperative templating, but after both senior surgeons agreed on the final stem size intraoperatively, C-arm fluoroscopy images were obtained with the last rasp size before stem implantation. The alignment and stem fitting of the femoral canal were evaluated. While evaluating the limb leg discrepancy anterior - posterior fluoroscopy image must include both hips and both lesser trochanters. Once this was achieved, the interteardrop line was used and vertical distance between interteardrop line and lesser trochanters measured for limb length discrepancy. Horizontal distance between tip of trochanter major and center of rotation was evaluated as lateral offset. For stem alignment, the femoral stem axis being parallel with the axis of the femoral canal was assessed. Also centralization of femoral stem tip in the femoral canal was assessed. Determination of stem was assessed according to full contact of broach teeth in sub trochanteric region. The stem was size changed unless all criteria above was achieved on fluoroscopy. After the operation, all patients were evaluated with X ray and CT(computerized tomography).

Medial canal flare index (MCFI) can be used for metaphyseal lacking femoral stems. The alignment of the femoral stem with the femoral canal, the limb length discrepancy ( LLD) and the lateral offsets were evaluated on X ray. The stem/endosteal areas at 2 cm above the trochanter minor (T+2) and 2 cm below the trochanter minor (T-2) and the deviation of the stem tip from the center of the femoral canal were evaluated on CT(Computerized tomography) images.

ELIGIBILITY:
Inclusion Criteria:

* patients with hip osteoarthritis

Exclusion Criteria:

* malignant tumors, previously known bone disease, drug consumption affecting bone mineralization or Crowe type III hip dislocations with greater than 4 cm of LLD were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
medial canal flare index ratios on computerized tomography images | 2 days after operation
  The stem/endosteal areas at 2 cm above the trochanter minor (T+2) and 2 cm below the trochanter minor (T-2) and the deviation of the stem tip from the center of the femoral canal were evaluated on CT images

SECONDARY OUTCOMES:
centralization of stem tip on computerized tomography images | 2 days after operation
  distance of stem tip from the center of medullary canal in millimeters
limb length discrepancy on X ray | 1 day after operation
  distance between interteardrop line to trochanter minor on anteroposterior x rays
lateral offset on Xray | 1 day after operation
  distance between trochanter major tip and hip's center of rotation
alignment of stem on computerized tomography | 2 days after operation
  the angle between axis of femoral canal and axis of stem

IPD SHARING:
Plan to Share IPD: Undecided